CLINICAL TRIAL: NCT07296952
Title: Using Implementation Science to Adapt a Targeted Transportation Intervention for Patients With Diabetic Retinopathy (PRONTO-EYE)
Acronym: PRONTO-EYE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Angel Scanzera, Associate Professor of Ophthalmology and Visual Sciences, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023-0960; K23EY034602 (NIH)
Record Dates: First submitted 2025-12-17; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Retinopathy (DR)
Keywords: diabetic retinopathy (DR); transportation; Medicaid
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Intervention Model Description: Hybrid Type 3 effectiveness-implemementation pilot feasibility trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRONTO-EYE rideshare intervention offered (Experimental): All eligible patients are invited to participate in PRONTO-EYE, a rideshare transportation program designed to improve adherence to eye care visits among Medicaid patients with diabetic retinopathy. All eligible patients are included in this arm regardless of if they decide to use PRONTO-EYE or not.
  Interventions: Behavioral: PRONTO-EYE

INTERVENTIONS:
Behavioral: PRONTO-EYE — The PROgram for Non-emergency TranspOrtation (PRONTO) - EYE intervention is a rideshare transportation program designed for patients to get to and from their visits. The intervention includes the rideshare as well as a service blueprint of the offering and how all individuals in the health system interact with it.

SUMMARY:
This is a a type 3 hybrid effectiveness-implementation pilot study to evaluate the PRONTO-EYE intervention, a rideshare transportation program, in patients with diabetic retinopathy with Medicaid insurance on adherence to ophthalmology visits.

DETAILED DESCRIPTION:
Vision loss is a public health issue that can limit every aspect of an individual's daily life, including communication, education, independence, mobility, and career goals. Diabetes is the leading cause of new cases of blindness in adults aged 18-64 years, with 1 in 8 adults with diabetes reporting severe visual difficulty or blindness in 2019. Though early detection and treatment can prevent visual impairment by as much as 90%, it is estimated that diabetic retinopathy (DR) is prevalent in 28.5-40.3% of the 37.3 million adults with diabetes in the U.S.

Because enhanced treatment options are available, prompt diagnosis and referral can improve visual outcomes and reduce complications, making adherence to visits critical. While DR treatment options have been shown to reduce complications and improve visual outcomes, barriers to eye care disproportionately affect under-resourced communities, resulting in underutilization of eye care services, delays in treatment, and poorer eye health outcomes.This research addresses a critical gap in our knowledge of how to identify patients with known DR and Medicaid insurance and provide a transportation intervention to get such individuals to needed eye care.

Using human-centered design methods, including qualitative interviews and workshops, journey mapping, and prototyping, investigators co-designed a rideshare intervention, PRONTO-EYE, to improve adherence to eye care visits in Medicaid patients with diabetic retinopathy. Upon completion of user testing, the service blueprint will be updated to meet key design criteria, including viability, feasibility, and desirability.

Investigators plan to conduct a type 3 hybrid effectiveness-implementation pilot study using a pre-post intervention design to evaluate the PRONTO-EYE intervention in Medicaid patients with diabetic retinopathy. Investigators will assess our primary outcome, adherence (defined as completing a scheduled ophthalmology visit), and secondary implementation outcomes, informed by the Proctor model, including acceptability, adoption, appropriateness, feasibility, fidelity, and penetration, through EHR data, surveys, and interviews. Our working hypothesis is that PRONTO-EYE will be successfully integrated into clinical workflows and increase adherence to visits compared to historical controls.

ELIGIBILITY:
Inclusion Criteria:

* Established patient
* Medicaid insurance
* History of diabetic retinopathy
* Lives within 25 miles of the clinic
* English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients that adhere to their scheduled ophthalmology visits | Baseline up to 6 months
  Proportion of patients who attend their scheduled ophthalmology visit compared to pre-implementation historical controls.

SECONDARY OUTCOMES:
Adoption of PRONTO-EYE | Assessed continuously throughout the up to 6-month feasibility trial, with a final summary at trial completion.
  Uptake and intention to employ the innovation, including percentage of patients who opt into rideshare and stakeholder buy-in, assessed via EHR data and interviews.
Appropriateness of PRONTO-EYE | Implementation outcomes will be assessed throughout the duration of the study
  Perceived fit, relevance, or compatibility of the intervention for the clinic's mission and patient needs, measured using questions adapted from the Intervention Appropriateness Measure (IAM) survey and interviews.
Feasibility of PRONTO-EYE | Assessed upon completion of the up to 6-month feasibility trial
  The number of rides successfully completed divided by the number of rides scheduled, as assessed via ride logs and observation.
Fidelity of PRONTO-EYE | Assessed continuously throughout the up to 6-month feasibility trial, with a final summary at trial completion.
  Degree to which the PRONTO-EYE transportation intervention was implemented as originally proposed, including adherence to planned processes for ride scheduling, patient eligibility criteria, and staff roles. Assessed via EHR data, program logs, and semi-structured interviews with staff.
Penetration of PRONTO-EyE | Assessed continuously throughout the up to 6-month feasibility trial, with a final summary at trial completion.
  Percentage of eligible patients using PRONTO-EYE among all eligible patients, assessed via EHR data.
Acceptability of PRONTO-EYE | Assessed continuously throughout the up to 6-month feasibility trial, with a final summary at trial completion.
  Perception among implementation stakeholders that the intervention is satisfactory, measured using questions adapted from the Acceptability of Intervention Measure (AIM) survey and semi-structured interviews.

IPD SHARING:
Plan to Share IPD: No
There are no plans to make IPD available to other researchers.